CLINICAL TRIAL: NCT00202124
Title: Double Blind Medium Term Efficacy Study of Trp01 in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Double Blind Study of Trp01 in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFW-TRP01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2002-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Tryptophan

INTERVENTIONS:
Drug: Tryptophan

SUMMARY:
The purpose of this study is to determine whether tryptophan is effective in the treatment of mild to moderate Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
The clinical trial will be a double-blind, placebo-controlled study with patients being randomized in a 2:1 ratio into groups A and B, respectively:

Group A: TRP01 1g b.i.d. for 26 weeks

Group B: placebo capsules b.i.d. for 26 weeks

After the initial screening, clinic visits will take place at 0, 13 and 26 weeks. The blinding will be maintained until all patients have completed the 26-week trial. Any patients wishing to continue taking the medication upon completion of the trial will be provided a prescription for the drug and may purchase it at their own expense.

ELIGIBILITY:
Inclusion Criteria:

Patients will be selected in order to fulfill both of the following definitions:

* Dementia according to DSM-IV criteria :

  * development of multiple cognitive deficits manifested by both memory impairment and one or more of the following cognitive disturbances: aphasia, apraxia, agnosia, disturbance in executive functioning
  * the above-mentioned deficits cause significant impairment in social or occupational functioning
  * they do not occur exclusively during the course of delirium
* Dementia according to communicative disorders and stroke criteria (NINCDS-ADRDA)

  * dementia established clinically and documented by a Folstein Mini-Mental State Examination (MMSE)
  * deficits in two or more areas of cognition
  * progressive worsening of memory and other cognitive functions
  * no disturbance of consciousness
  * absence of systematic disorders or other brain diseases that in and of themselves can account for progressive deficit in memory and cognition

Furthermore, patients must fulfill the following criteria:

* men, or postmenopausal or surgically sterilized women
* with severity of dementia of mild to moderate degree as reflected by a score of greater than 14 but less than 26 on the MMSE
* with a minimum one-year duration of the symptomatology (progressive worsening of memory and other cognitive functions)
* living at home or in an institution provided that they have reliable caregivers
* able to perform the required psychometric tests and evaluations. Visual and auditory acuity (with glasses or hearing aid if required) must be sufficient to complete the protocol-specified procedures.
* Clinical laboratory battery (see section 7.2.2) must yield results within normal limits or determined as not clinically significant by the study physician for the patient's sex and age
* Patients and their substitute decision-makers must have signed the written informed consent form

Exclusion Criteria:

Patients with any of the following will not be included in the study:

* Patients with any other cause of dementia as evidenced by medical history, general physical and neurological examination, laboratory tests, and neuroradiological findings:

  * Vascular dementia, as evidenced by Modified Hachinski Ischemia Scale
  * Depressive pseudementia, as evidenced by cognitive disturbances concomitant to a major depressive episode according to DSM-IV and/or a history of more than one major depressive episode
  * DSM-IV criteria for any major psychiatric disorder including schizophrenia, alcohol or substance abuse
  * Huntington's chorea or Parkinson's disease, evidenced by neurological examination, with an onset prior to or concurrent with dementia
  * Creutzfeldt-Jakob disease
  * Intracranial mass lesion
  * Clinically important head injury
  * History or current evidence of stroke
  * Onset of dementia following cardiac arrest or heart surgery
  * Neurosyphilis
  * Seropositivity for HIV
  * Vitamin B12 deficiency
  * Uncorrected hypothyroidism (i.e. abnormal free T4, ultrasensitive TSH)
* Patients with other relevant concomitant diseases:

  * Patients with history or current evidence of a sleep disorder
  * Patients with a clinically significant cardiovascular, renal, hepatic, pulmonary, gastrointestinal, endocrine, metabolic, opthalmologic, or hematologic condition
  * Current evidence or history within the past year of myocardial infarction (MI), congestive heart failure
  * Blood pressure at screening of > 180 mm Hg systolic or 100 mm Hg diastolic
  * Impaired renal, hepatic, or gastrointestinal function, which could interfere with drug absorption, metabolism or excretion
  * Seizure disorder
  * Diabetes
  * Earlier diagnosis or current evidence of cataracts
  * Progressive fatal disease (other than AD)
  * Treatment with any other investigational drug in the last 8 weeks prior to screening
  * Previous administration of TRP01

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12
Dates: Start 2001-04; Study Completion 2002-03

PRIMARY OUTCOMES:
1. MMSE score
2. Alzheimer's Disease Assessment Scale, cognitive subpart (ADAS-Cog) as an evaluation of cognitive functioning

SECONDARY OUTCOMES:
1. Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC)
2. Neuropsychiatric Inventory (NPI)
3. Disability Assessment for Dementia (DAD)
4. Physical Self-Maintenance Scale (PSMS)
5. Functional Activities Questionnaire (FAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Donald F Weaver, MD, PhD, Study Chair — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada